CLINICAL TRIAL: NCT01227824
Title: A Randomized, Double Blind Study of the Safety and Efficacy of GSK1349572 50mg Once Daily to Raltegravir 400mg Twice Daily Both Administered With Fixed-dose Dual Nucleoside Reverse Transcriptase Inhibitor Therapy Over 96 Weeks in HIV-1 Infected Antiretroviral Therapy Naive Adult Subjects
Brief Title: A Trial Comparing GSK1349572 50mg Once Daily to Raltegravir 400mg Twice Daily
Acronym: SPRING-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113086
Record Dates: First submitted 2010-10-14; First posted 2010-10-25 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: integrase inhibitor; HIV Infection; raltegravir; GSK1349572
MeSH Terms: conditions — Infections; HIV Infections | interventions — dolutegravir; Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1349572 (N=~394) (Experimental): GSK1349572 50mg once daily + raltegravir placebo twice daily + NRTI background therapy once daily
  Interventions: Drug: GSK1349572 (dolutegravir); Other: GSK1349572 Placebo; Other: ABC/3TC; Other: TDF/FTC
- raltegravir (N=~394) (Active Comparator): raltegravir 400mg twice daily + GSK1349572 placebo once daily + NRTI background therapy once daily
  Interventions: Drug: raltegravir; Other: ABC/3TC; Other: TDF/FTC; Other: raltegravir Placebo

INTERVENTIONS:
Drug: GSK1349572 (dolutegravir) — GSK1349572 50 mg taken once daily with or without food
  Arms: GSK1349572 (N=~394)
Drug: raltegravir — raltegravir 400mg taken twice daily
  Arms: raltegravir (N=~394)
Other: GSK1349572 Placebo — GSK1349572 placebo taken once daily
  Arms: GSK1349572 (N=~394)
Other: ABC/3TC — Abacavir/Lamivudine background therapy once daily
Other: TDF/FTC — Tenofovir/emtricitabine background therapy once daily
Other: raltegravir Placebo — raltegravir placebo taken twice daily
  Arms: raltegravir (N=~394)

SUMMARY:
The purpose of this trial is to assess the non-inferior antiviral activity of GSK1349572 50 mg once daily versus RAL 400mg twice daily over 48 weeks; non-inferiority will also be tested at Week 96. Both GSK1349572 and RAL will be given in combination with fixed-dose dual NRTI therapy (ABC/3TC or TDF/FTC). This study will be conducted in HIV-1 infected ART-naïve adult subjects.

DETAILED DESCRIPTION:
ING113086 is a Phase 3 randomized, double-blind, double dummy, active-controlled, multicenter, study conducted in approximately 788 HIV-1 infected ART-naïve subjects. Subjects will be randomized 1:1 one of the following treatment arms:

1. GSK1349572 50 mg once daily (approximately 394 subjects) + fixed-dose dual NRTI therapy (either ABC/3TC or TDF/FTC)

   OR
2. 400 mg RAL twice daily (approximately 394 subjects) + fixed-dose dual NRTI therapy (either ABC/3TC or TDF/FTC)

Analyses will be conducted at 48 weeks and 96 weeks. Subjects randomized to receive GSK1349572 and who successfully complete 96 weeks of treatment will continue to have access to GSK1349572 through the study until either it is locally available, as long as they continue to derive clinical benefit.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Screening plasma HIV-1 RNA ≥1000 c/mL
* Antiretroviral-naïve (≤ 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection)
* Ability to understand and sign a written informed consent form
* Willingness to use approved methods of contraception to avoid pregnancy (women of child bearing potential only)
* Age equal to or greater than 18 years

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Active Center for Disease and Prevention Control (CDC) Category C disease
* Moderate to severe hepatic impairment
* Anticipated need for HCV therapy during the study
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Malignancy within the past 5 years
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents or any immunomodulator within 28 days of Screening
* Exposure to an agent with documented activity against HIV-1 in vitro or an experimental vaccine or drug within 28 days of first dose of study medication
* Primary viral resistance in the Screening result
* Verified Grade 4 laboratory abnormality
* ALT >5 xULN
* ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin);
* Estimated creatinine clearance <50 mL/min
* Recent history (≤3 months) of upper or lower gastrointestinal bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2010-10-19; Primary Completion 2012-02-06 (Actual); Study Completion 2016-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (81):
- United States (18):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Surry Hills, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (9):
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (6):
  - GSK Investigational Site, Cona (Ferrara), Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Rovigo, Veneto
- Russia (10):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, N.Novgorod
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Volgograd
- Spain (19):
  - GSK Investigational Site, (Móstoles) Madrid
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo ( Pontevedra)
- United Kingdom (4):
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Crumpsall, Manchester
  - GSK Investigational Site, London

REFERENCES:
- [Background] Brinson C, Walmsley S, Arasteh K, et al. Dolutegravir treatment response and safety by key subgroups in treatment naive HIV-infected individuals. Published at: Conference on Retroviruses and Opportunistic Infections - 20th Annual; March 3-6, 2013; Atlanta, GA.
- [Background] Raffi F, Rachlis A, Stellbrink HJ, Hardy WD, Torti C, Orkin C, Bloch M, Podzamczer D, Pokrovsky V, Pulido F, Almond S, Margolis D, Brennan C, Min S; SPRING-2 Study Group. Once-daily dolutegravir versus raltegravir in antiretroviral-naive adults with HIV-1 infection: 48 week results from the randomised, double-blind, non-inferiority SPRING-2 study. Lancet. 2013 Mar 2;381(9868):735-43. doi: 10.1016/S0140-6736(12)61853-4. Epub 2013 Jan 8. PMID 23306000
- [Derived] Raffi F, Jaeger H, Quiros-Roldan E, Albrecht H, Belonosova E, Gatell JM, Baril JG, Domingo P, Brennan C, Almond S, Min S; extended SPRING-2 Study Group. Once-daily dolutegravir versus twice-daily raltegravir in antiretroviral-naive adults with HIV-1 infection (SPRING-2 study): 96 week results from a randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2013 Nov;13(11):927-35. doi: 10.1016/S1473-3099(13)70257-3. Epub 2013 Sep 25. PMID 24074642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, parallel group, non-inferiority study to demonstrate the antiviral activity of Dolutegravir. Participants were enrolled from 9 countries. Participants in Dolutegravir arm who completed 96 Weeks double-blind phase continued to receive Dolutegravir in open-label phase, until dolutegravir was locally available commercially.
Pre-assignment Details: Total 1035 participants were screened; 827 participants were randomized, and 822 participants entered the treatment period. Of the 5 participants who were randomized but not treated with investigational product, 4 withdrew consent and 1 was randomized in error. 338 participants were enrolled in open label phase to receive Dolutegravir.
Groups:
- DTG 50 mg Once a Day: Participants received Dolutegravir (DTG) 50 milligrams (mg) once a day in combination with Nonnucleoside Reverse Transcriptase Inhibitor (NRTI) therapy, either with Abacavir (ABC)/Lamivudine (3TC) or Tenofovir (TDF)/Emtricitabine (FTC). Participants were given the opportunity to receive DTG 50 mg once a day during an Open-label Phase of the study.
- RTG 400 mg BID: Participants received Raltegravir (RTG) 400 mg twice a day (BID) in combination with NRTI therapy, either with ABC/3TC or TDF/FTC.
- DTG 50 mg Once a Day (Open-label): Participants who successfully completed 96 weeks of double blind phase continued to receive DTG 50 mg once a day during open label phase, until dolutegravir was locally available commercially. Participants received DTG 50 mg once a day in combination with NRTI therapy, with either ABC/3TC or TDF/FTC.
Period: Double-blind Phase: 96 Weeks Duration
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID | DTG 50 mg Once a Day (Open-label)
Started | 411 | 411 | 0
Completed | 304 | 332 | 0
Not Completed | 107 | 79 | 0
Not completed — Adverse Event | 12 | 7 | 0
Not completed — Lack of Efficacy | 22 | 25 | 0
Not completed — Protocol Violation | 18 | 16 | 0
Not completed — Met Protocol-defined Stopping Criteria | 6 | 3 | 0
Not completed — Study Closed/Terminated | 6 | 4 | 0
Not completed — Lost to Follow-up | 22 | 10 | 0
Not completed — Withdrawal by Subject | 18 | 14 | 0
Not completed — Physician Decision | 3 | 0 | 0
Period: Open-label Phase: Median of 1267 Days
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID | DTG 50 mg Once a Day (Open-label)
Started | 0 | 0 | 338 (338 participants continued into the Open-label phase on completing the Double-blind Phase)
Completed | 0 | 0 | 294
Not Completed | 0 | 0 | 44
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 5
Not completed — Protocol Violation | 0 | 0 | 5
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 8
Not completed — Physician Decision | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- DTG 50 mg Once a Day: Participants received DTG 50 mg once a day in combination with NRTI therapy, either with ABC/3TC or TDF)/FTC. Participants were given the opportunity to receive DTG 50 mg once a day during an Open-label Phase of the study.
- RTG 400 mg BID: Participants received RTG 400 mg BID in combination with NRTI therapy, either with ABC/3TC or TDF/FTC.
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID | Total
Number analyzed (Participants) | 411 | 411 | 822
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (9.19) | 36.6 (10.02) | 37.0 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 56 | 119
  Male | 348 | 355 | 703
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage (Her) | 49 | 39 | 88
  American Indian or Alaska Native | 7 | 9 | 16
  Central/South Asian Her | 2 | 0 | 2
  Japanese/East Asian Her/South East Asian Her | 4 | 10 | 14
  Native Hawaiian or other Pacific Islander | 2 | 0 | 2
  White | 346 | 352 | 698
  African American/African Her and Asian and White | 1 | 0 | 1
  Asian and White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) [HIV-1RNA] <50 Copies (c)/Milliliter (mL) Through Week 48
Description: Percentage of participants with plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) with <50 c/mL was assessed using the Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) snapshot algorithm. The algorithm treats all participants without HIV-1 RNA data as non-responders, as well as participants who switch their concomitant Antiretroviral Therapy (ART) prior to Week 48 as follows: background ART substitutions not permitted per study; background ART substitutions permitted per study unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure will be determined by the last available HIV-1 RNA assessment while the subject was on-treatment. Intent-to-Treat Exposed (ITT-E) Population comprised all randomized participants who received at least one dose of study medication.
Time Frame: Baseline up to Week 48
Population: ITT-E Population.
Measure: Number; unit: Percentage of participants
Groups:
- DTG 50 mg Once a Day: Participants received DTG 50 mg once a day in combination with NRTI therapy, either with ABC/3TC or TDF/FTC. Participants were given the opportunity to receive DTG 50 mg once a day during an Open-label Phase of the study.
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Percentage of participants | 88 | 85
Statistical Analysis 1: Comparison: DTG 50 mg Once a Day vs RTG 400 mg BID; Test type: Non-Inferiority or Equivalence — Non-inferiority could be concluded if the lower bound of a two-sided 95% confidence interval for the difference (DTG - RAL) in percentages between the two treatment arms was > -10%; Difference in percentage = 2.5, 95% CI 2-sided [-2.2 to 7.1] — Analysis was based on Cochran-Mantel Haenszel stratified analysis adjusted for the following Baseline stratification factors: baseline HIV-1 RNA and background dual NRTI

2. Secondary Outcome: Number of Participants With Detectable HIV-1 Virus That Has Genotypic or Phenotypic Evidence of INI Resistance.
Description: Number of participants with detectable virus that has genotypic or phenotypic evidence of Integrase Inhibitor (INI) resistance were assessed at Week 48 and Week 96. Integrase inhibitors are a class of antiretroviral drug designed to block the action of integrase, a viral enzyme that inserts the viral genome into the deoxyribonucleic acid (DNA) of the host cell.
Time Frame: Week 48 and Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Participants
  Week 48, genotypic | 0 | 1
  Week 48, phenotypic | 1 | 2
  Week 96, genotypic | 0 | 1
  Week 96, phenotypic | 1 | 2

3. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL
Description: The number of participants with plasma HIV-1 RNA level <50 c/mL was assessed at Week 96.
Time Frame: Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Participants | 332 | 314

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <400 c/mL
Description: The number of participants with plasma HIV-1 RNA level <400 c/mL was assessed at Week 48 and Week 96.
Time Frame: Week 48 and Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Participants
  Week 48 | 369 | 356
  Week 96 | 338 | 321

5. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA Over Time
Description: Change from Baseline in plasma HIV-1 RNA over time was assessed at Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96. Baseline was defined as the measurements performed on Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96
Population: ITT-E Population.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
log10 c/mL
  Baseline n=411, 411 | 4.538 (0.7258) | 4.599 (0.7048)
  Week 4, n=402, 406: number analyzed (Participants) | 402 | 406
  Week 4, n=402, 406 | -2.817 (0.6198) | -2.801 (0.6041)
  Week 8, n=397, 402: number analyzed (Participants) | 397 | 402
  Week 8, n=397, 402 | -2.897 (0.6837) | -2.886 (0.6754)
  Week 12, n=396, 395: number analyzed (Participants) | 396 | 395
  Week 12, n=396, 395 | -2.908 (0.6863) | -2.918 (0.6834)
  Week 16, n=395, 388: number analyzed (Participants) | 395 | 388
  Week 16, n=395, 388 | -2.917 (0.6949) | -2.943 (0.6841)
  Week 24, n=393, 390: number analyzed (Participants) | 393 | 390
  Week 24, n=393, 390 | -2.896 (0.7889) | -2.933 (0.7398)
  Week 32, n=386, 377: number analyzed (Participants) | 386 | 377
  Week 32, n=386, 377 | -2.907 (0.7609) | -2.947 (0.7613)
  Week 40, n=375, 358: number analyzed (Participants) | 375 | 358
  Week 40, n=375, 358 | -2.920 (0.7219) | -2.946 (0.6700)
  Week 48, n=374, 358: number analyzed (Participants) | 374 | 358
  Week 48, n=374, 358 | -2.915 (0.7237) | -2.942 (0.6737)
  Week 60, n=366, 355: number analyzed (Participants) | 366 | 355
  Week 60, n=366, 355 | -2.912 (0.7344) | -2.937 (0.6685)
  Week 72, n=361, 350: number analyzed (Participants) | 361 | 350
  Week 72, n=361, 350 | -2.917 (0.7261) | -2.932 (0.6728)
  Week 84, n=352, 338: number analyzed (Participants) | 352 | 338
  Week 84, n=352, 338 | -2.932 (0.7073) | -2.916 (0.6646)
  Week 96, n=342, 329: number analyzed (Participants) | 342 | 329
  Week 96, n=342, 329 | -2.938 (0.7004) | -2.901 (0.7072)

6. Secondary Outcome: Absolute Values in Plasma HIV-1 RNA Over Time
Description: Absolute values in plasma HIV-1 RNA over time was assessed at Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96. Only those participants with data available at the specified time points were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96
Population: ITT-E Population.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
log10 c/mL
  Baseline n=411, 411 | 4.538 (0.7258) | 4.599 (0.7048)
  Week 4, n=402, 406: number analyzed (Participants) | 402 | 406
  Week 4, n=402, 406 | 1.718 (0.2593) | 1.800 (0.4095)
  Week 8, n=397, 402: number analyzed (Participants) | 397 | 402
  Week 8, n=397, 402 | 1.646 (0.2006) | 1.709 (0.3791)
  Week 12, n=396, 395: number analyzed (Participants) | 396 | 395
  Week 12, n=396, 395 | 1.626 (0.1323) | 1.672 (0.3125)
  Week 16, n=395, 388: number analyzed (Participants) | 395 | 388
  Week 16, n=395, 388 | 1.620 (0.1252) | 1.648 (0.2647)
  Week 24, n=393, 390: number analyzed (Participants) | 393 | 390
  Week 24, n=393, 390 | 1.643 (0.2950) | 1.655 (0.3476)
  Week 32, n=386, 377: number analyzed (Participants) | 386 | 377
  Week 32, n=386, 377 | 1.620 (0.1917) | 1.636 (0.2721)
  Week 40, n=375, 358: number analyzed (Participants) | 375 | 358
  Week 40, n=375, 358 | 1.603 (0.0821) | 1.601 (0.0784)
  Week 48, n=374, 358: number analyzed (Participants) | 374 | 358
  Week 48, n=374, 358 | 1.606 (0.0866) | 1.599 (0.0582)
  Week 60, n=366, 355: number analyzed (Participants) | 366 | 355
  Week 60, n=366, 355 | 1.605 (0.1134) | 1.599 (0.0560)
  Week 72, n=361, 350: number analyzed (Participants) | 361 | 350
  Week 72, n=361, 350 | 1.601 (0.0803) | 1.605 (0.0836)
  Week 84, n=352, 338: number analyzed (Participants) | 352 | 338
  Week 84, n=352, 338 | 1.607 (0.1337) | 1.614 (0.1279)
  Week 96, n=342, 329: number analyzed (Participants) | 342 | 329
  Week 96, n=342, 329 | 1.599 (0.830) | 1.630 (0.2515)

7. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD)4+ Cell Counts Over Time
Description: CD4 lymphocyte cells (also called T-cells or T-helper cells) are the primary targets of HIV. The CD4 count and the CD4 percentage mark the degree of immuno compromise. The CD4 count is used to stage the participants disease, determine the risk of opportunistic illnesses, assess prognosis, and guide decisions about when to start ART. Changes from Baseline in CD4+ cell counts over time was assessed at Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96. Baseline was defined as measurements performed on Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96
Population: ITT-E Population.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Cells per cubic millimeter (cells/mm^3)
  Baseline n=411, 411 | 379.2 (178.32) | 374.3 (163.37)
  Week 4, n=398, 403: number analyzed (Participants) | 398 | 403
  Week 4, n=398, 403 | 93.3 (116.27) | 97.2 (129.35)
  Week 8, n=398, 402: number analyzed (Participants) | 398 | 402
  Week 8, n=398, 402 | 121.6 (127.97) | 126.6 (134.59)
  Week 12, n=392, 397: number analyzed (Participants) | 392 | 397
  Week 12, n=392, 397 | 130.7 (131.49) | 145.1 (144.08)
  Week 16, n=394, 392: number analyzed (Participants) | 394 | 392
  Week 16, n=394, 392 | 155.1 (137.23) | 173.0 (159.10)
  Week 24, n=392, 389: number analyzed (Participants) | 392 | 389
  Week 24, n=392, 389 | 199.3 (161.23) | 204.2 (162.28)
  Week 32, n=384, 375: number analyzed (Participants) | 384 | 375
  Week 32, n=384, 375 | 223.4 (165.30) | 241.3 (167.64)
  Week 40, n=371, 357: number analyzed (Participants) | 371 | 357
  Week 40, n=371, 357 | 224.1 (173.59) | 239.8 (173.33)
  Week 48, n=374, 357: number analyzed (Participants) | 374 | 357
  Week 48, n=374, 357 | 238.9 (171.81) | 257.5 (178.69)
  Week 60, n=367, 355: number analyzed (Participants) | 367 | 355
  Week 60, n=367, 355 | 247.8 (184.11) | 264.2 (188.63)
  Week 72, n=360, 350: number analyzed (Participants) | 360 | 350
  Week 72, n=360, 350 | 247.8 (168.37) | 278.6 (182.76)
  Week 84, n=351, 338: number analyzed (Participants) | 351 | 338
  Week 84, n=351, 338 | 281.3 (175.07) | 292.9 (199.42)
  Week 96, n=343, 328: number analyzed (Participants) | 343 | 328
  Week 96, n=343, 328 | 292.2 (195.70) | 286.2 (192.45)

8. Secondary Outcome: Absolute Values in CD4+ Cell Counts Over Time
Description: CD4 lymphocyte cells (also called T-cells or T-helper cells) are the primary targets of HIV. The CD4 count and the CD4 percentage mark the degree of immuno compromise. The CD4 count is used to stage the patient's disease, determine the risk of opportunistic illnesses, assess prognosis, and guide decisions about when to start antiretroviral therapy absolute values in CD4+ cell counts over time was assessed at Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96. Only those participants with data available at the specified time points were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96
Population: ITT-E Population.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
cells/mm^3
  Baseline n=411, 411 | 379.2 (172.32) | 374.3 (163.37)
  Week 4, n=398, 403: number analyzed (Participants) | 398 | 403
  Week 4, n=398, 403 | 474.2 (199.06) | 471.8 (191.02)
  Week 8, n=398, 402: number analyzed (Participants) | 398 | 402
  Week 8, n=398, 402 | 502.3 (205.15) | 502.4 (187.99)
  Week 12, n=392, 397: number analyzed (Participants) | 392 | 397
  Week 12, n=392, 397 | 513.3 (218.75) | 518.3 (195.59)
  Week 16, n=394, 392: number analyzed (Participants) | 394 | 392
  Week 16, n=394, 392 | 536.4 (219.47) | 550.1 (221.77)
  Week 24, n=392, 389: number analyzed (Participants) | 392 | 389
  Week 24, n=392, 389 | 582.0 (232.93) | 580.8 (218.76)
  Week 32, n=384, 375: number analyzed (Participants) | 384 | 375
  Week 32, n=384, 375 | 606.5 (242.95) | 618.7 (237.56)
  Week 40, n=371, 357: number analyzed (Participants) | 371 | 357
  Week 40, n=371, 357 | 609.1 (239.11) | 623.1 (234.82)
  Week 48, n=374, 357: number analyzed (Participants) | 374 | 357
  Week 48, n=374, 357 | 623.8 (247.82) | 641.2 (241.75)
  Week 60, n=367, 355: number analyzed (Participants) | 367 | 355
  Week 60, n=367, 355 | 635.6 (241.27) | 648.5 (238.99)
  Week 72, n=360, 350: number analyzed (Participants) | 360 | 350
  Week 72, n=360, 350 | 635.2 (237.78) | 664.0 (239.86)
  Week 84, n=351, 338: number analyzed (Participants) | 351 | 338
  Week 84, n=351, 338 | 668.0 (246.50) | 677.5 (249.64)
  Week 96, n=343, 328: number analyzed (Participants) | 343 | 328
  Week 96, n=343, 328 | 679.8 (257.89) | 672.4 (237.54)

9. Secondary Outcome: Number of Participants With the Indicated Post-Baseline HIV-associated Conditions and Progression, Excluding Recurrences
Description: Clinical disease progression (CDP) was assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the AIDS surveillance case definition. Indicators of CDP were defined as: CDC CAT A at Baseline to a CDC CAT C event (EV); CDC CAT B at Baseline to a CDC CAT C EV; CDC CAT C at Baseline to a new CDC CAT C EV; or CDC CAT A, B, or C at Baseline to death.
Time Frame: From Baseline until Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Participants
  Any category condition | 10 | 8
  Any Category B condition | 3 | 3
  Any Category C condition | 6 | 4
  Any death | 1 | 1
  Progression from CAT A to CAT C | 4 | 2
  Progression from CAT B to CAT C | 3 | 1
  Progression from CAT C to new CAT C | 0 | 1
  Progression from CAT A, B, or C to death | 1 | 1

10. Secondary Outcome: Number of Participants With the Indicated Grade 1 to 4 Clinical Chemistry and Hematology Toxicities/Laboratory Adverse Events (AEs)
Description: All Grade 1 to 4 post-Baseline-emergent chemistry toxicities included alanine aminotransferase (ALT), alkaline phosphatase (ALP), asparate aminotransferase (AST), carbon dioxide (CO2) content/bicarbonate, cholesterol, creatine kinase (CK), creatinine, hyperglycemia, hyperkalemia, hypernatremia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) cholesterol calculation, lipase, phosphorus inorganic, total bilirubin, and triglycerides. All Grade 1 to 4 post-Baseline-emergent hematology toxities included hemoglobin, platelet count, total neutrophils, and white blood cell count. The Division of AIDS (DAIDS) defined toxicity grades as follows: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening; Grade 5, death. Safety Population: all participants who received at least one dose of investigational product
Time Frame: From Baseline until Week 96
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 411 | 411
Participants
  ALT | 57 | 70
  ALP | 7 | 15
  AST | 67 | 75
  CO2 content/bicarbonate | 58 | 67
  Cholesterol | 90 | 73
  CK | 61 | 47
  Creatinine | 11 | 7
  Hyperglycaemia | 70 | 87
  Hyperkalemia | 7 | 4
  Hypernatremia | 4 | 6
  Hypoglycaemia | 17 | 27
  Hypokalemia | 10 | 15
  Hyponatremia | 34 | 48
  LDL cholesterol calculation | 74 | 49
  Lipase | 55 | 62
  Phosphorus, inorganic | 65 | 71
  Total bilirubin | 27 | 24
  Triglycerides | 7 | 8
  Hemoglobin | 10 | 5
  Platelet count | 19 | 19
  Total neutrophils | 54 | 48
  White Blood Cell count | 19 | 7

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time Tau [AUC(0-tau)] of DTG
Description: AUC is defined as the area under the DTG concentration-time curve as a measure of drug exposure over time. AUC(0-tau) is defined as the area under the plasma concentration-time curve from time zero to time tau over a dosing interval at steady state, where tau is the length of the dosing interval of DTG. The predicted individual AUC(0-tau) were obtained from the final population PK model by an empirical Bayes estimation. Blood samples for PK assessments were collected at pre-dose (within 15 minutes prior to dose) at Week 4, Week 24, and Week 48 and 1 to 3 hours post-dose or 4 to 12 hours post-dose at Week 4 and Week 24. If 1 to 3 hours post-dose was completed at Week 4, then the 4 to12 hour post-dose must be obtained at Week 48, and vice versa. The Pharmacokinetic (PK) Concentration Population comprised of all participants who received DTG, had undergone PK sampling during the study, and provided evaluable DTG plasma concentration data.
Time Frame: Week 4, Week 24, and Week 48
Population: PK Concentration Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter(µg*hr/mL)
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 403 | 0
Micrograms*hour per milliliter(µg*hr/mL) | 53.6 (26.8) |

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) and Concentration at the End of a Dosing Interval (Ctau) of DTG
Description: The maximum plasma concentration (Cmax) and concentration at the end of a dosing interval (Ctau) of DTG were assessed at Week 48. The predicted individual Cmax and Ctau were obtained from the final population PK model by simulation of the concentration-time profiles. Blood samples for PK assessments were collected at pre-dose (within 15 minutes prior to dose) at Week 4, Week 24, and Week 48 and 1 to 3 hours post-dose or 4 to 12 hours post-dose at Week 4 and Week 24. If 1 to 3 hour post-dose was completed at Week 4, then the 4 to12 hour post-dose must be obtained at Week 48, and vice versa.
Time Frame: Week 4, Week 24, and Week 48
Population: PK Concentration Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | DTG 50 mg Once a Day | RTG 400 mg BID
Number analyzed (Participants) | 403 | 0
Micrograms per milliliter (µg/mL)
  Cmax | 3.69 (19.6) |
  Ctau | 1.10 (46.5) |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the study (up to a median of 1267 days).
Description: AEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Groups:
- RTG 400mg BID: Participants received RTG 400 mg BID in combination with NRTI therapy, either with ABC/3TC or TDF/FTC.
- DTG 50 mg Once a Day (Open-label): Participants who successfully completed 96 weeks of double blind phase continued to receive DTG 50 mg once a day during open label phase, until DTG was locally available commercially. Participants received DTG 50 mg once a day in combination with NRTI therapy, with either ABC/3TC or TDF/FTC.
Arm/Group | DTG 50 mg Once a Day | RTG 400mg BID | DTG 50 mg Once a Day (Open-label)
All-Cause Mortality (participants affected / at risk) | 1/411 | 1/411 | 0/338
Serious Adverse Events (participants affected / at risk) | 41/411 | 45/411 | 21/338
Other Adverse Events (participants affected / at risk) | 353/411 | 344/411 | 256/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 50 mg Once a Day (N=411) | RTG 400mg BID (N=411) | DTG 50 mg Once a Day (Open-label) (N=338)
Appendicitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 3 (4) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Homicide (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Keratoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Polyserositis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 50 mg Once a Day (N=411) | RTG 400mg BID (N=411) | DTG 50 mg Once a Day (Open-label) (N=338)
Diarrhoea (Gastrointestinal disorders) | 58 (72) | 54 (65) | 21 (25)
Viral upper respiratory tract infection (Infections and infestations) | 54 (73) | 54 (77) | 24 (27)
Headache (Nervous system disorders) | 56 (63) | 55 (70) | 9 (9)
Nausea (Gastrointestinal disorders) | 60 (70) | 55 (66) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 34 (43) | 31 (38) | 27 (36)
Syphilis (Infections and infestations) | 24 (25) | 28 (30) | 24 (30)
Bronchitis (Infections and infestations) | 24 (33) | 22 (25) | 15 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (27) | 26 (29) | 10 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 22 (24) | 9 (9)
Fatigue (General disorders) | 22 (26) | 24 (27) | 7 (7)
Insomnia (Psychiatric disorders) | 28 (28) | 19 (20) | 6 (6)
Pyrexia (General disorders) | 23 (30) | 24 (26) | 6 (7)
Sinusitis (Infections and infestations) | 25 (36) | 16 (18) | 12 (19)
Depression (Psychiatric disorders) | 26 (26) | 18 (18) | 8 (8)
Dizziness (Nervous system disorders) | 24 (25) | 24 (24) | 0 (0)
Anxiety (Psychiatric disorders) | 19 (19) | 22 (24) | 6 (7)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (17) | 22 (24) | 8 (9)
Gastroenteritis (Infections and infestations) | 18 (21) | 18 (23) | 10 (11)
Pharyngitis (Infections and infestations) | 23 (31) | 14 (16) | 9 (9)
Influenza (Infections and infestations) | 16 (17) | 22 (23) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 18 (21) | 16 (20) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 16 (19) | 6 (7)
Asthenia (General disorders) | 14 (16) | 18 (19) | 7 (7)
Vomiting (Gastrointestinal disorders) | 16 (21) | 18 (19) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 18 (22) | 19 (23) | 1 (1)
Respiratory tract infection (Infections and infestations) | 19 (19) | 12 (14) | 5 (9)
Rhinitis (Infections and infestations) | 13 (20) | 13 (15) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 14 (17) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (18) | 10 (10) | 5 (5)
Constipation (Gastrointestinal disorders) | 15 (16) | 14 (17) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 12 (13) | 12 (14) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 15 (15) | 9 (9) | 5 (6)
Influenza like illness (General disorders) | 13 (15) | 9 (11) | 7 (8)
Oral herpes (Infections and infestations) | 8 (9) | 13 (17) | 7 (8)
Conjunctivitis (Infections and infestations) | 8 (8) | 11 (11) | 8 (9)
Flatulence (Gastrointestinal disorders) | 12 (12) | 11 (11) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 12 (12) | 5 (6)
Urinary tract infection (Infections and infestations) | 12 (14) | 7 (8) | 4 (4)
Abnormal dreams (Psychiatric disorders) | 13 (14) | 8 (9) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 11 (13) | 7 (8) | 4 (6)
Urethritis (Infections and infestations) | 9 (10) | 8 (10) | 5 (6)
Chlamydial infection (Infections and infestations) | 5 (6) | 9 (13) | 7 (8)
Gonorrhoea (Infections and infestations) | 7 (8) | 6 (7) | 8 (9)
Tendonitis (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9) | 5 (5)
Herpes zoster (Infections and infestations) | 9 (9) | 9 (9) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7) | 3 (3)
Seasonal allergy (Immune system disorders) | 8 (8) | 7 (7) | 5 (7)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 7 (7)
Acne (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (9) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 11 (11) | 2 (3)
Gingivitis (Infections and infestations) | 8 (8) | 11 (11) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 8 (10) | 2 (2)
Tonsillitis (Infections and infestations) | 10 (10) | 4 (4) | 5 (8)
Folliculitis (Infections and infestations) | 6 (7) | 8 (9) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (11) | 1 (1)
Toothache (Gastrointestinal disorders) | 9 (10) | 3 (3) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 12 (12) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) | 6 (8)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 6 (7) | 4 (5)
Ear infection (Infections and infestations) | 7 (7) | 7 (11) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 9 (13) | 4 (4) | 3 (4)
Sleep disorder (Psychiatric disorders) | 7 (7) | 8 (8) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 8 (9) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 7 (9) | 7 (10) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8) | 2 (2)
Sciatica (Nervous system disorders) | 4 (4) | 7 (9) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (5) | 6 (6) | 3 (3)
Genital herpes (Infections and infestations) | 5 (6) | 4 (5) | 5 (6)
Libido decreased (Psychiatric disorders) | 3 (3) | 10 (10) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 5 (5)
Pneumonia (Infections and infestations) | 8 (8) | 4 (4) | 2 (2)
Proctitis (Gastrointestinal disorders) | 5 (5) | 5 (6) | 4 (4)
Tooth infection (Infections and infestations) | 7 (8) | 4 (4) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (4) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 7 (7) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (7) | 4 (4) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (13) | 0 (0)
Secondary syphilis (Infections and infestations) | 4 (4) | 4 (5) | 5 (5)
Anogenital dysplasia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 5 (5) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 10 (11) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (8) | 4 (10) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (2)
Cellulitis (Infections and infestations) | 5 (5) | 4 (5) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 7 (8) | 3 (5)
Herpes virus infection (Infections and infestations) | 3 (3) | 5 (8) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (8) | 2 (2)
Onychomycosis (Infections and infestations) | 4 (5) | 4 (4) | 3 (3)
Chest pain (General disorders) | 5 (5) | 2 (2) | 3 (3)
Fungal skin infection (Infections and infestations) | 5 (5) | 5 (5) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 3 (3)
Migraine (Nervous system disorders) | 4 (5) | 5 (10) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 2 (2)
Stress (Psychiatric disorders) | 4 (4) | 4 (4) | 2 (2)
Urethritis gonococcal (Infections and infestations) | 2 (2) | 5 (5) | 3 (3)
Viral infection (Infections and infestations) | 6 (6) | 4 (4) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3) | 4 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 4 (9) | 2 (2)
Furuncle (Infections and infestations) | 3 (3) | 4 (5) | 2 (2)
Lethargy (Nervous system disorders) | 3 (3) | 6 (7) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 5 (7) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 4 (5) | 0 (0)
Tooth abscess (Infections and infestations) | 4 (4) | 3 (3) | 2 (3)
Weight increased (Investigations) | 4 (4) | 5 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (5) | 4 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 2 (2) | 2 (2)
Nightmare (Psychiatric disorders) | 6 (6) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)
Tinea infection (Infections and infestations) | 5 (5) | 3 (3) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 3 (3)
Lymphogranuloma venereum (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Otitis media (Infections and infestations) | 4 (4) | 2 (4) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 1 (1)
Tinea versicolour (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 5 (5) | 0 (0)
Weight decreased (Investigations) | 3 (4) | 3 (3) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1)
Blood pressure increased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 5 (6) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0)
Urethral discharge (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 2 (3) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Disturbance in attention (Nervous system disorders) | 1 (1) | 4 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Erysipelas (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Facial paralysis (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (5) | 1 (1)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Labyrinthitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Proctitis gonococcal (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Amnesia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Drug use disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Feeling abnormal (General disorders) | 2 (3) | 2 (2) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 3 (3) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5)
Intertrigo (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (4)
Malaise (General disorders) | 3 (3) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Orchitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 2 (4) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 1 (2)
Acute hepatitis C (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Balanitis candida (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Burnout syndrome (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 3 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Epididymitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Giardiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 2 (4) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Local swelling (General disorders) | 3 (3) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Parotitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pilonidal cyst (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Primary syphilis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urethral pain (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Angular cheilitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Cyst (General disorders) | 2 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatophytosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Facial wasting (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis shigella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Genital infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Granuloma (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 2 (2)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Infection parasitic (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Mucosal dryness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oesophageal spasm (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Urinary sediment present (Investigations) | 0 (0) | 2 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acne conglobata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agnosia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agoraphobia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood testosterone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body fat disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicitis human papilloma virus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Circadian rhythm sleep disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Epididymal tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heart sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Human papilloma virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypospermia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ichthyosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jarisch-Herxheimer reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Kidney duplex (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Lactase deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Latent syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lip haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental fatigue (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema mucosal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oestradiol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Palatal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Panic reaction (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papilloma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parasite stool test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phobia of flying (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Proctitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
QRS axis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Shigella test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep-related eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Spider naevus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Stress at work (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sycosis barbae (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testis discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thymus disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vaginitis gardnerella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Yersinia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.